CLINICAL TRIAL: NCT04318717
Title: Adjuvant Pembrolizumab and Hypofractionated Radiation Therapy for the Treatment of Mucosal Melanoma
Brief Title: Pembrolizumab and Hypofractionated Radiation Therapy for the Treatment of Mucosal Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202003124
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Mucosal Melanoma of the Head and Neck
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Pembrolizumab + Hypofractionated radiation therapy (Experimental): * Pembrolizumab will be given intravenously over 30 minutes (-5/+10 minutes) at a dose of 200 mg on an outpatient basis on Day 1 of each 21-day cycle for a total of up to 12 months (17 cycles).
  * Hypofractionated radiation therapy may be given at any point during the first 2 cycles of pembrolizuimab. It should begin within 90 days of surgical resection. Intensity modulated radiation therapy (IMRT) or intensity modulated proton therapy (IMPT) are to be used exclusively. IMRT or IMPT will be delivered twice per week in five fractions of 6 Gy given over 2.5 weeks totaling 30 Gy.
  Interventions: Drug: Pembrolizumab; Radiation: Hypofractionated radiation therapy

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is commercially available
  Other Names: Keytruda
Radiation: Hypofractionated radiation therapy — It is preferred to leave at least 48 hours between fractions. Daily imaging to verify accurate set-up is mandatory.

SUMMARY:
This is an open-label, single center, one cohort, non-randomized, phase II study. The aim is to evaluate the efficacy and safety of the combination of hypofractionated radiotherapy (HRT) and pembrolizumab on local tumor control in mucosal melanoma patients. Treatment effect will be compared with historical radiation therapy-alone control data.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed mucosal melanoma that has undergone surgical resection. Patient must not have received prior radiation therapy within the area of interest.
* At least 16 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 70%)
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,200/mcL
  * Platelets ≥ 100,000/mcL
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (IULN)
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine clearance > 30 mL/min by Cockcroft-Gault
* The effects of pembrolizumab on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry, for the duration of study participation, and 6 months after last dose of pembrolizumab. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of the study, and 6 months after last dose of pembrolizumab.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* A history of other malignancy with the exception of malignancies for which all treatment was completed at least 2 years before registration and the patient has no evidence of disease.
* Received radiation therapy within the area of interest.
* Currently receiving any other investigational agents.
* Metastatic disease.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment. The use of up to 10 mg/day of prednisone or equivalent is approved and does not exclude the patient from the trial.
* Active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, > 10 mg of prednisone per day, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. The use of up to 10 mg/day of prednisone or equivalent is approved and does not exclude the patient from the trial.
* Has a history of (non-infectious) pneumonitis/Interstitial lung disease that required maintenance steroids (>10 mg of prednisone) or current pneumonitis/interstitial lung disease.
* Has received a live vaccine or live-attenuated vaccination within 30 days of planned treatment start. Administration of killed vaccines is allowed.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2020-05-29 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2032-07-31 (Estimated)

PRIMARY OUTCOMES:
Local tumor control rate | 1 year after completion of treatment (estimated to be 2 years)
  Tumor control rate is defined as the percentage of subjects at 12 months who are free of local recurrence, regional recurrence, distant recurrence, second primary cancer, or death.

SECONDARY OUTCOMES:
Number of treatment-related grade 3 or greater adverse events | Baseline through 90 days after end of treatment (estimated to be 15 months)
  The total number of adverse events determined to be treatment related and grade 3 or higher as assessed using CTCAE v5.0 criteria.
Number of treatment discontinuations due to treatment-related adverse events | Through end of treatment (estimated to be 1 year)
  The total number of participants who discontinued treatment due to treatment-related adverse events as assessed using CTCAE v5.0 criteria.
Relapse-free survival (RFS) | At 3 years after completion of treatment (estimated to be 4 years)
  -Defined as the duration of time from the start date of study treatment to the date of earliest disease relapse or death, whichever occurs first. Patients who neither relapse nor die by the data cutoff date will be censored at the last follow up date.
Distant metastasis-free survival | At 3 years after completion of treatment (estimated to be 4 years)
  -Defined as the duration of time from the start date of study treatment to the date of appearance of a distant metastasis or death, whichever occurs first. Patients who neither develop distant metastasis nor die by the data cutoff date will be censored at the last follow up date.
Overall survival | At 3 years after completion of treatment (estimated to be 4 years)
  -Defined as the duration of time from the start date of study treatment to death from any cause. Patients who are alive by the data cutoff date will be censored at the last follow up date.

CONTACTS AND LOCATIONS:
Overall Officials: George Ansstas, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu